CLINICAL TRIAL: NCT01451255
Title: Early Detection of Pulmonary Arterial Hypertension Using Cardiac Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian Shapiro, Principal Investigator, Mayo Clinic
Other Study IDs: 11-002576
Record Dates: First submitted 2011-10-08; First posted 2011-10-13 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension
Keywords: pulsatility; normal subjects; mild pulmonary hypertension; exercise-associated pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Cardiac magnetic resonance imaging has emerged as a potential valuable test for the early detection of Pulmonary Arterial Hypertension. A number of reports have provided some preliminary evidence that Pulmonary Artery (PA) stiffness may be accurately detected by imaging of the pulmonary artery in order to measure PA stiffness. In addition, cardiac MRI could play provide early and effective treatment for Pulmonary Arterial Hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients aged ≥ 18 years with PAH as dictated by a comprehensive examination and echocardiography will be included for enrollment.

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Mechanical ventilation
* Acute or chronic renal failure (creatinine clearance < 30 ml/min or requiring renal replacement therapy)
* Inability to perform MRI (i.e. claustrophobia, severe obesity (> 150 kg), device incompatible with MRI)
* Significant arrhythmia that precludes adequate ECG-gating for the MRI (i.e. atrial fibrillation with highly variable cycle lengths)
* Prior heart or lung transplantation
* Left ventricular systolic (ejection fraction < 50%) or diastolic failure (based on Framingham criteria for heart failure with preserved ejection fraction)
* Significant left-sided valvular disease (≥ moderate aortic stenosis, mitral stenosis, aortic regurgitation, mitral regurgitation) or prior valve surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will consist of a total of 90 subjects separated evenly into the following subgroups: 1) Mild PAH, 2) Moderate or Severe PAH, and 3) Normal Controls.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Shapiro, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida

REFERENCES:
- [Derived] Ray JC, Burger C, Mergo P, Safford R, Blackshear J, Austin C, Fairweather D, Heckman MG, Zeiger T, Dubin M, Shapiro B. Pulmonary arterial stiffness assessed by cardiovascular magnetic resonance imaging is a predictor of mild pulmonary arterial hypertension. Int J Cardiovasc Imaging. 2019 Oct;35(10):1881-1892. doi: 10.1007/s10554-018-1397-y. Epub 2018 Jun 22. PMID 29934885